CLINICAL TRIAL: NCT01834898
Title: Phase 4 Study, Open, Observational, to Evaluate the Safety and Tolerability of Hydrochloride Controlled-release Oxycodone in Moderate and Severe Postoperative Pain in Oncologic Head and Neck Surgery.
Brief Title: Safety and Tolerability of Controlled-release Oxycodone on Postoperative Pain in Oncologic Head and Neck Surgery
Status: Completed | Type: Observational
Sponsor: Instituto Nacional de Cancer, Brazil (Other Government)
Responsible Party: Sponsor
Other Study IDs: INCA 10/2010; IncaBrazil (Other: Instituto Nacional de Câncer)
Record Dates: First submitted 2013-04-10; First posted 2013-04-18 (Estimated); Last update posted 2013-04-18 (Estimated); Status verified 2013-04

CONDITIONS: Postoperative Nausea; Adverse Effects; Opioid Analgesic Adverse Reaction; Pain
Keywords: postoperative; analgesia; adverse effects; opioid; oxycodone
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Pain; Agnosia | interventions — Analgesics, Opioid

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Controlled-release oxycodone: Controlled-released oxycodone. First day postoperatively, 40 mg / day divided into 20 mg of 12 in 12 hours and in the second postoperative day, 20 mg / day divided into 10 mg of 12 in 12 hours
  Interventions: Drug: Controlled-release oxycodone

INTERVENTIONS:
Drug: Controlled-release oxycodone — Controlled-release oxycodone. First day postoperatively, 40 mg / day divided into 20 mg of 12 in 12 hours and in the second postoperative day, 20 mg / day divided into 10 mg of 12 in 12 hours
  Other Names: Opioid; Postoperative analgesia; Postoperative pain

SUMMARY:
The hypothesis of this study is that controlled release oxycodone can be safe and well tolerated for the control of postoperative pain in surgery for head and neck cancer. The primary objective is to study the safety and the incidence and severity of adverse effects, and the secondary objective is to evaluate the analgesic efficacy and identify the frequency of use of rescue medication and the prescribing physician's opinion about the quality of postoperative analgesia with oxycodone controlled release in oncologic surgery of the head and neck.

DETAILED DESCRIPTION:
Phase IV clinical trial, observational, prospective, open approved by the Research Ethics Committee of the National Cancer Institute José Alencar Gomes da Silva - INCA, Brazil (no. 10/2010). The Instrument of Consent is signed by all patients.

Eighty-three patients will be included. Ages between 18 and 70 years both genders, 2 and 3 American Society of Anesthesiologists physical status, which present moderate to severe pain source postoperative surgical oncology, head and neck, medium and large, elective, non-emergency, able to swallow tablets whole (not chewed, broken or crushed) in the immediate postoperative period after recovery of cognitive functions. Will be excluded pregnant or breastfeeding, allergic to oxycodone and other opioids, gastrectomized or colostomized, asthmatics with severe organ dysfunction, with a history or suspected paralytic ileus, or a history psychiatric disorders, severe respiratory depression, patients who are receiving opioid analgesics in baseline, history of abuse of alcohol and illicit drugs, patients who present in plasma glutamic oxaloacetic transaminase above 48 U / l (men) and 40 U / I (women) and / or glutamic pyruvic transaminase above 53 U / l (men) and 40 U / I (women) and patients who present plasma creatinine above 1.7 mg / dl and / or urea above 65 mg / dl. All patients will be assessed preoperatively seven to one day before surgery (visit 1) when will the signed consent form, proceeded to pre-anesthetic evaluation and blood will be collected for laboratory tests: complete blood count, β-human chorionic gonadotropin(women), glutamic oxaloacetic transaminase, glutamic pyruvic transaminase, creatinine and urea.

In the immediate postoperative period (visit 2), the pain will be assessed by verbal numeric scale (VNS) and when pain is moderate to severe (≥ 4 EVN) and the patient is lucid and able to swallow, will start orally controlled-release oxycodone (Oxycontin, Zodiac Pharmaceuticals, Brazil) at a dose of 20 mg (tablets whole without crushing or division), administered by the investigator. Every 12 hours and a subsequent period of 48 hours after the first dose of oxycodone controlled-release, the pain will be evaluated again, and the occurrence and intensity of adverse events (visits 3, 4, 5 and 6 respectively 12 , 24, 36 and 48 hours after the first dose of oxycodone). The doses of controlled-release oxycodone will be standardized as follows: on the first day postoperatively, 40 mg / day divided into 20 mg of 12 in 12 hours and in the second postoperative day, 20 mg / day divided into 10 mg of 12 in 12 hours.

The rescue medication will be used non opioids analgesics as paracetamol, dipyrone, diclofenac or tenoxicam, only after the first administration of controlled-release oxycodone postoperatively. During the visits described above will be annotated to rescue analgesia and its frequency, should it ever be used between doses of oxycodone.

Between post-operative 7 and 13 days will be held the visit 7, which will be evaluated pain intensity (EVN), the occurrence and severity of adverse effects, and the investigator's opinion about treatment. Finally, the patient's blood will be collected to perform the same tests listed at visit 1, except β-human chorionic gonadotropin (women), and the study was terminated.

Sample Size and Statistical Analysis

When considering the occurrence of nausea of 25% as a safety parameter, assessed by literature data, the number of patients required will be 72. Taking into consideration a dropout of about 20% will require 86 patients in total (to an accuracy of 10%, around the percentage confidence interval (CI) 95%). The study of normal age variable will be conducted with the test Kolmogorov - Smirnov. The Friedman test is used to compare medians of pain intensity from visit 2 to visit 7. The Dunn test will be used for post-hoc comparisons (between two) of median pain intensity (p <0.001 - significant). The McNemar test for pairwise comparisons of proportions will be employed for comparisons of adverse events (visits 4, 5, 6 and 7 with respect to visit 3) (p <0.05 = significant). The remaining data will be presented by frequency.

ELIGIBILITY:
Inclusion Criteria:

* patients on postoperative head and neck oncologic surgery
* 2 and 3 American Society of Anesthesiologists physical status
* moderate to severe postoperative pain
* elective surgery
* able to swallow tablets whole (not chewed, broken or crushed) in the immediate postoperative period after recovery of cognitive functions.

Exclusion Criteria:

* pregnant or breastfeeding
* allergic to oxycodone and other opioids
* gastrectomized or colostomized
* asthmatics with severe organ dysfunction
* history or suspected paralytic ileus
* history psychiatric disorders
* severe respiratory depression
* patients who are receiving opioid analgesics in baseline
* history of abuse of alcohol and illicit drugs
* plasma glutamic oxaloacetic transaminase above 48 U / l (men) and 40 U / I (women) and / or glutamic pyruvic transaminase above 53 U / l (men) and 40 U / I (women)
* plasma creatinine above 1.7 mg / dl and / or urea above 65 mg / dl
* emergency surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients on postoperative head and neck oncologic surgery which moderate to severe pain
Sampling Method: Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2010-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with nausea | 48 hours post dose
  number of participants with nausea 48 hours after first dose of controlled-released oxycodone

SECONDARY OUTCOMES:
Pain intensity | 48 hours post dose
  pain intensity by numerical scale 48 hours after the first dose of controlled released oxycodone

OTHER OUTCOMES:
Degree of quality of postoperative analgesia | At the seventh postoperative day
  Investigator's opinion about treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ismar L Cavalcanti, MD PhD, Principal Investigator — Instituto Nacional de Câncer Brazil
Locations (1):
- Instituto Nacional de Câncer José Alencar Gomes da Silva, Rio de Janeiro, Rio de Janeiro, Brazil